CLINICAL TRIAL: NCT02495363
Title: Analgesic Effects of Ultrasound Guided PEC Blocks on Analgesic Opioid Consumption of Cancer Surgery Patients
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 201-15
Record Dates: First submitted 2015-06-18; First posted 2015-07-13 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2016-10

CONDITIONS: Malignant Neoplasm of Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PECS block in additions to general anesthesia: As standard analgesic protocol participants undergoing mastectomy surgeries under general anesthesia will have an addition of Pectoral Block regional anesthesia.
  Following obtaining written informed consent, ultrasound guided PECS Block will be performed by identifying the thoracic muscles, in addition to general anesthesia Following the identification, the investigator will inject the anesthetic solution which will contain the conventional 25 cc of Bupivacaine 0.25-0.5% .
  Interventions: Procedure: PECS Block; Drug: Bupivacaine 0.25-0.5%

INTERVENTIONS:
Procedure: PECS Block — As standard departmental protocol ultrasound guided PECS Block will be performed by identifying the thoracic muscles. Following the identification, the investigator will inject the anesthetic solution which will contain the conventional 25 cc of Bupivacaine 0.25-0.5% .
  The concentration is determined by the upper dose limit to 2 mg / kg 11
Drug: Bupivacaine 0.25-0.5% — Ultrasound guided PECS Block will be performed by identifying the thoracic muscles. Following the identification, the investigator will inject the anesthetic solution which will contain the conventional 25 cc of Bupivacaine 0.25-0.5% .
  The concentration is determined by the upper dose limit to 2 mg / kg 11

SUMMARY:
Examining the analgesic effect of ultrasound guided Pectoral Blocks on analgesic opioid consumption after surgical removal of breast tissue.

This study's uniqueness is in the quantification of the analgesic effect of regional anesthesia on its influence to reduce the use of opioid substances, and the variety of side effects associated with them, which has yet to been described in literature.

DETAILED DESCRIPTION:
This is a prospective, observational,single center study which will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital. Sixty women undergoing breast tissue resection under general anesthesia will be enrolled after filling out an informed consent form.

As standard protocol in our hospital all participants will include women undergoing the surgery under general anesthesia, and the an addition of regional PEC block anesthesia.

The use of opioid substances during surgery will be done under the discretion of the anesthesiologist, according to accepted professional criteria.

All participants will undergo the the PEC block before surgery under general anesthesia under aseptic conditions, which is the standard analgesia protocol in our department.

Ultrasound guided PECS Block will be performed by identifying the thoracic muscles. Following the identification, the investigator will inject the anesthetic solution which will contain the conventional 25 cc of Bupivacaine 0.25-0.5% .

The concentration is determined by the upper dose limit to 2 mg / kg 11.

At the end of the operation all participants will be transferred to the post anesthesia recovery supervision unit, as standard protocol. The women will receive analgesic treatment according to accepted recovery unit protocols of Beilinson Hospital, and according to the professional discretion of the anesthesiologist in charge of the recovery unit.

On postoperative day one all participants will be asked to fill out a questionnaire that measures the degree of their pain after surgery, and the extent of the expected side effects from exposure to opioids This questionnaire is based on a questionnaire measuring quality QoR recovery from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Women over 18 who undergo breast tissue resection under general anesthesia at Beilinson Hospital, and are able to comply with the study's protocol

Exclusion Criteria:

1. Lack of patient's consent or lack of patient's ability to provide consent.
2. Known hypersensitivity to local anesthetic or to opioid, which will affect the nature of the pain management therapy in these patients.
3. Existing evidence of infection or gangrene on the thorax which prevents implementation of regional anesthesia - .
4. Known coagulation disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women above 18 undergoing breast tissue resection under general anesthesia at Beilinson Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scales quantification of the analgesic effect of PECS Block regional anesthesia on its influence to reduce the use of opioid substances, and the variety of side effects associated with them | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petach Tikvah, Israel

REFERENCES:
- [Background] Poleshuck EL, Katz J, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for chronic pain following breast cancer surgery: a prospective study. J Pain. 2006 Sep;7(9):626-34. doi: 10.1016/j.jpain.2006.02.007. PMID 16942948
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Background] Power I. An update on analgesics. Br J Anaesth. 2011 Jul;107(1):19-24. doi: 10.1093/bja/aer126. Epub 2011 May 30. PMID 21624966
- [Background] Fujii Y. Management of postoperative nausea and vomiting in women scheduled for breast cancer surgery. J Anesth. 2011 Dec;25(6):917-22. doi: 10.1007/s00540-011-1241-1. Epub 2011 Oct 1. PMID 21964679 (Retraction: PMID 23455701 Hirota K. J Anesth. 2013 Apr;27(2):322)
- [Background] Shin SW, Cho AR, Lee HJ, Kim HJ, Byeon GJ, Yoon JW, Kim KH, Kwon JY. Maintenance anaesthetics during remifentanil-based anaesthesia might affect postoperative pain control after breast cancer surgery. Br J Anaesth. 2010 Nov;105(5):661-7. doi: 10.1093/bja/aeq257. Epub 2010 Sep 28. PMID 20876698
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Abdallah FW, Morgan PJ, Cil T, McNaught A, Escallon JM, Semple JL, Wu W, Chan VW. Ultrasound-guided multilevel paravertebral blocks and total intravenous anesthesia improve the quality of recovery after ambulatory breast tumor resection. Anesthesiology. 2014 Mar;120(3):703-13. doi: 10.1097/ALN.0000436117.52143.bc. PMID 24071616
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540